CLINICAL TRIAL: NCT07084506
Title: RETROSPECTIVE COLLECTION OF SAFETY AND PERFORMANCE DATA
Brief Title: RETROSPECTIVE COLLECTION OF SAFETY AND PERFORMANCE DATA - 2023.02
Status: Completed | Type: Observational
Sponsor: Bioceramed (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023.02
Record Dates: First submitted 2025-06-05; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Bone Defects; Dental Area

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study, based on observations of clinical practice, aims to collect clinical data to update information on the performance and safety of the n-IBS® when used according to its intended purpose and current clinical applications. The results of the clinical study will serve as clinical evidence to support the assessment of the device's safety and performance, contributing to the overall clinical evaluation of the product.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females (aged > 18 years old);
* Patients who were implanted with the synthetic bone substitute n-IBS® for the treatment of intrabony defects associated with periodontal disease or for bone augmentation procedures in the alveolar process and maxillary sinus regions.

Exclusion Criteria:

* Patients with infection at the implantation site;
* Patients with metabolic disorders affecting bone healing;
* Patients with immune system disorders;
* Patients with systemic conditions that impair bone healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged > 18 years old) undergoing reconstructive dental surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Performance Endpoint | follow-up visits, through study completion, an average of 1 year
  Assessment of bone consolidation at the surgical site, based on the quantification of bone gain (mm) as measured through routine X-ray imaging, to evaluate osseous regeneration.
2. Safety Endpoint | Follow-up visits, through study completion, an average of 1 year
  Assessment of Adverse Events (AEs) related to n-IBS® during the follow-up period of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Center Cabinet Dentaire de Stomatologie & Implantologie, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No